CLINICAL TRIAL: NCT02536469
Title: A Phase Ib, Dose Escalation, Multiple Dose Trial With HuMax-IL8 in Patients With Metastatic or Unresectable, Locally Advanced Malignant Solid Tumors
Brief Title: HuMax-IL8 (Interleukin8) in Patients With Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: This trial was conducted previously by Cormorant (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COR01CD101; CA027-001 (Other: BMS)
Record Dates: First submitted 2015-08-23; First posted 2015-08-31 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Solid Tumor
MeSH Terms: interventions — HuMax-IL8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HuMax-IL8 (Experimental): HuMax-IL8 drug product intended for intravenous infusion. Subjects will be treated every 2 weeks. Every 2 doses (4 weeks) will be considered 1 cycle
  Interventions: Drug: HuMax-IL8

INTERVENTIONS:
Drug: HuMax-IL8 — HuMax-IL8 drug product intended for intravenous infusion. Subjects will be treated every 2 weeks. Every 2 doses (4 weeks) will be considered 1 cycle
  Other Names: BMS-968253

SUMMARY:
A phase Ib, dose escalation, multiple dose trial with HuMax-IL8 in patients with metastatic or unresectable, locally advanced malignant solid tumors.

DETAILED DESCRIPTION:
All human subjects with a diagnosis of incurable solid tumors are eligible for the dose-escalation phase of this study. This study consists of two phases, the dose-escalation phase and the expansion phase. Subjects will be treated with the study treatment until any off-treatment criteria are met. The safety and efficacy will be assessed until the end of treatment or for a maximum of 52 weeks. In addition, a separate visit will be performed at the time of disease progression if the patient has a progression between end of treatment and 52 weeks. The patients will be followed up for overall survival until the study closure. The study will be closed when all enrolled patients have been followed up for at least 52 weeks or have died.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have metastatic or unresectable locally advanced malignant solid tumor.
* Patients may have measurable or non-measurable but evaluable disease.
* Patients with surgically resected metastatic disease at high risk of relapse are also eligible.
* Patients must have completed or had disease progression on at least one prior line of disease-appropriate therapy for metastatic disease, or not be candidates for therapy of proven efficacy for their disease.
* Patients must have recovered (grade 1 or baseline) from any clinically significant toxicity associated with prior therapy
* Age ≥ 18 years. .
* ECOG (Eastern Cooperative Oncology Group) performance status ≤ 1 (Karnofsky ≥ 70%).
* Patients must have normal organ and hematologic function therapy
* Patients must have baseline pulse oximetry > 90% on room air

Exclusion Criteria:

* Pregnant women or women presently breast-feeding
* Concurrent treatment for cancer
* Chronic hepatitis B or C infection.
* Any significant disease that, in the opinion of the investigator, may impair the patient's tolerance of study treatment.
* Significant dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Active autoimmune diseases requiring treatment or a history of autoimmune disease.
* Concurrent use of systemic steroids
* Patients who are receiving any other investigational agents
* Patients with untreated central nervous system metastases or local treatment of brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the agent used in study.
* Serious or uncontrolled intercurrent illness
* HIV-positive patients are ineligible
* Patients unwilling to use adequate contraception

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who experience DLTs (Dose Limiting Toxicity) 28 days following the first dose of HuMax-IL8, as well as all DLTs occurring during the study thereafter. | From cycle 1 day 1 up to 28 days
  The primary endpoint of this study is the proportion of patients who experience DLTs. The MTD (Maximum Tolerated Dose) will be determined based on the dose escalation cohorts. The evaluation period for DLTs will be 28 days following the first dose of HuMax-IL8

SECONDARY OUTCOMES:
Pharmacokinetic properties of HuMax-IL8 in patients including AUC (Area Under the Curve) | From baseline up to 72 hours after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- National Cancer Institute, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Bilusic M, Heery CR, Collins JM, Donahue RN, Palena C, Madan RA, Karzai F, Marte JL, Strauss J, Gatti-Mays ME, Schlom J, Gulley JL. Phase I trial of HuMax-IL8 (BMS-986253), an anti-IL-8 monoclonal antibody, in patients with metastatic or unresectable solid tumors. J Immunother Cancer. 2019 Sep 5;7(1):240. doi: 10.1186/s40425-019-0706-x. PMID 31488216
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx